CLINICAL TRIAL: NCT01762150
Title: Sorafenib Combined With Cisplatin and Gemcitabine for the Treatment of Patients With Advanced Renal Collecting Duct Carcinoma:A Pilot, Open Study
Brief Title: Sorafenib Combined With Chemotherapy for Renal Collecting Duct Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Jun Guo, Director of renal cancer and melanoma department, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCH-RCC-120601
Record Dates: First submitted 2012-12-22; First posted 2013-01-07 (Estimated); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Renal Cell Carcinoma
Keywords: collected duct carcinoma; sorafenib
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sorafenib; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- sorafenib combined with chemotherapy (Experimental): this trial is designed single arm. all the subjects enrolled will receive the experimental intervention,ie. sorafenib+gemcitabine+cisplatin.
  Interventions: Drug: Sorafenib; Drug: Gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Drug: Sorafenib — Sorafenib 400mg BID by oral until progressed;
  Other Names: Nexavar
Drug: Gemcitabine — Gemcitabine: 1000mg/m2, administered by intravenous drip for 30~60min on Day 1 and 8,for 4 cycles;
  Other Names: Gemzar
Drug: Cisplatin — Cisplatin: 25mg/m2, administered by intravenous drip on Day 1-3, with appropriate liquid hydration,for 4 cycles.
  Other Names: Cis-Dichlorodiamineplatinum

SUMMARY:
The goal of this clinical research study is to learn the effectiveness of sorafenib combined with gemcitabine plus cisplatin in the treatment of patients with locally advanced or metastatic collecting duct carcinoma(CDC) of the kidney. The safety of each treatment will also be studied.

DETAILED DESCRIPTION:
Collecting duct carcinoma(CDC) of the kidney is a rare and aggressive neoplasm of the distal collecting tubules for which there is no established treatment. Since the histology of collecting duct carcinoma is similar to that of urothelial carcinoma, a prospective phase II trial in France(2007) studied gemcitabine plus cisplatin as the first-line treatment of advanced CDC, resulting an effective rate of 26%. The targeted drugs can produce definite efficacy on renal clear cell carcinoma, but the data on targeted drugs for the treatment of renal advanced collecting duct carcinoma is limited. We sponsored this study based on the assumption that targeted drugs combined with chemotherapy can produce additive, positive effects in CDC.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years, ≤70 years, male or female;
* Advanced collecting duct carcinoma of the kidney is diagnosed histologically or pathologically ;
* Have not received anti-angiogenesis targeted drug therapy and systemic chemotherapy;
* Have at least one measurable tumor lesion (Response Evaluation Criteria In Solid Tumors);
* Eastern Cooperative Oncology Group（ECOG) performance scale is 0 or 1;
* The expected life span is ≥12 weeks;
* No contraindications for chemotherapy, with enough liver function and renal function and normal ECG recording.Peripheral hemogram: neutrophil≥1.5×109/L, Plt≥100×109/L, Hgb≥90 g/L;Renal function: serum creatinine≤1.5 folds the upper limit of normal (ULN); For patients with non-metastatic liver dysfunction: alanine aminotransferase and aspartate aminotransferase≤2.5 ULN, For patients with metastatic liver dysfunction: alanine aminotransferase and aspartate aminotransferase≤5 ULN;
* The patients participate voluntarily and have signed the informed consent form.

Exclusion Criteria:

* Pregnant and lactating women, or female patients of child-bearing age without taking contraceptive measures;
* Patients with severe acute infection without being controlled effectively or having pyogenic and chronic infections with persistently unhealed wounds;
* Past history of serious heart diseases, including: cardiac function classification ≥NYHA class II, unstable angina pectoris, myocardial infarction, arrhythmia requiring anti-arrhythmic drug therapy (excluding β-blockers or digoxin), and uncontrolled hypertension;
* Patients with a history of HIV infection or active phase of chronic hepatitis B/C;
* negative imaging examination result 4 weeks prior to enrollment);
* Epilepsy patients requiring drug therapy (e.g. steroids or antiepileptic drugs);
* A history of allogeneic organ transplantation;
* Patients with evidence of hemorrhagic constitution or a past history of hemorrhage;
* Patients currently receiving renal dialysis;
* Past or present concomitant tumors with the primary lesions or histological characteristics different from the tumors evaluated in this study, excluding other tumor cured longer than 3 years before enrollment;
* Patients participating in other clinical trials simultaneously;
* Other conditions unsatisfying the inclusion criteria in the investigator's opinions.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-06; Primary Completion 2016-12 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
progress-free survival,PFS | Time from enrollment to the dates of disease progression,death from any cause or last tumor assessment reported between date of first patient enrollment until 30 June 2015 cut of date
  Progression Free Survival is defined as the time from enrollment to the date of first documented disease progression or death from any cause.

SECONDARY OUTCOMES:
adverse event, AE | Time from enrollment to the dates of disease progression,death from any cause or last tumor assessment reported between date of first patient enrollment until 30 June 2015 cut of date
  Any events,no matter related to interventions,occur during the period from the enrollment to death or 30 days after withdrawal from the trial

OTHER OUTCOMES:
objective response rate (ORR) | Time from enrollment to the dates of disease progression,death from any cause or last tumor assessment reported between date of first patient enrollment until 30 June 2015 cut of date
  CR:complete response PR:partial response ORR:CR+PR
overall survival (OS) | Time from enrollment to the dates of death from any cause or last follow up reported between date of first patient enrollment until 30 June 2015 cut of date
  Time from enrollment to the dates of death from any cause or last follow up reported between date of first patient enrollment until 30 June 2015 cut of date
the rate of progress-free survive | Time from enrollment to the dates of disease progression,death from any cause or last tumor assessment reported between date of first patient enrollment until 30 June 2015 cut of date
  the proportion of patients who don't experience progress at 3,6,9 months after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Jun Guo, MD,PHD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (5):
- China (5):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Sun Yat-sen university cancer center, Guangzhou, Guangdong
  - Shenyang general hospital of Shenyang military command, Shenyang, Liaoning
  - Xijing Hospital, Xi’an, Shanxi
  - West China Hospital, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Oudard S, Banu E, Vieillefond A, Fournier L, Priou F, Medioni J, Banu A, Duclos B, Rolland F, Escudier B, Arakelyan N, Culine S; GETUG (Groupe d'Etudes des Tumeurs Uro-Genitales). Prospective multicenter phase II study of gemcitabine plus platinum salt for metastatic collecting duct carcinoma: results of a GETUG (Groupe d'Etudes des Tumeurs Uro-Genitales) study. J Urol. 2007 May;177(5):1698-702. doi: 10.1016/j.juro.2007.01.063. PMID 17437788
- [Background] Escudier B, Eisen T, Stadler WM, Szczylik C, Oudard S, Siebels M, Negrier S, Chevreau C, Solska E, Desai AA, Rolland F, Demkow T, Hutson TE, Gore M, Freeman S, Schwartz B, Shan M, Simantov R, Bukowski RM; TARGET Study Group. Sorafenib in advanced clear-cell renal-cell carcinoma. N Engl J Med. 2007 Jan 11;356(2):125-34. doi: 10.1056/NEJMoa060655. PMID 17215530
- [Derived] Sheng X, Cao D, Yuan J, Zhou F, Wei Q, Xie X, Cui C, Chi Z, Si L, Li S, Mao L, Lian B, Tang B, Yan X, Wang X, Kong Y, Dai J, Bai X, Zhou L, Guo J. Sorafenib in combination with gemcitabine plus cisplatin chemotherapy in metastatic renal collecting duct carcinoma: A prospective, multicentre, single-arm, phase 2 study. Eur J Cancer. 2018 Sep;100:1-7. doi: 10.1016/j.ejca.2018.04.007. Epub 2018 Jun 19. PMID 29933095